CLINICAL TRIAL: NCT00000373
Title: Neurobiology/Treatment of Obsessive-Compulsive Disorder
Brief Title: Treatment of Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH045802 (NIH); R01MH045802 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Adolescence; Adult; Antipsychotic Agents; Dopamine Antagonists; Female; Fluvoxamine; Haloperidol; Human; Male; Middle Age; Obsessive-Compulsive Disorder; Placebos; Serotonin Uptake Inhibitors; Tourette Syndrome; Tryptophan; Drug Combinations; Antipsychotic Agents -- *therapeutic use; Fluvoxamine -- *therapeutic use; Haloperidol -- *therapeutic use; Obsessive-Compulsive Disorder -- *drug therapy; Obsessive-Compulsive Disorder -- physiopathology; Serotonin Uptake Inhibitors -- *therapeutic use
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Tourette Syndrome | interventions — olanzapine-fluoxetine combination; Fluoxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- olanzapine + fluoxetine (Active Comparator): The specific aim was to determine whether combined treatment with fluoxetine plus olanzapine would be more effective than fluoxetine plus placebo in treating OCD subjects who were partial or nonresponders to a prospective, 8-week, open-label trial of fluoxetine.
  Interventions: Drug: placebo + fluoxetine
- placebo + fluoxetine (Placebo Comparator): The specific aim was to determine whether combined treatment with fluoxetine plus olanzapine would be more effective than fluoxetine plus placebo in treating OCD subjects who were partial or nonresponders to a prospective, 8-week, open-label trial of fluoxetine.
  Interventions: Drug: olanzapine + fluoxetine

INTERVENTIONS:
Drug: olanzapine + fluoxetine
  Arms: placebo + fluoxetine
Drug: placebo + fluoxetine
  Arms: olanzapine + fluoxetine

SUMMARY:
The purpose of this study is to find the best treatment for Tourette's Syndrome (TS)-spectrum obsessive-compulsive disorder (OCD), which includes symptoms of TS, e.g., repeated and involuntary body movements (tics).

There are 2 parts to this study: In Part 1, patients are placed into 1 of 2 groups based on type of OCD, determined by medical history and family member interviews. In Part 2, patients are treated with fluvoxamine (FVX) for 8 weeks. If patients do not respond to FVX alone, either haloperidol or an inactive placebo will be added to the FVX regimen; patients will take this drug combination for 4 weeks. Patients will be monitored throughout the trial.

DETAILED DESCRIPTION:
To advance the neurobiology and treatment of obsessive-compulsive disorder (OCD) by focusing on Tourette's Syndrome (TS)-spectrum OCD as a possible homogeneous form of OCD, and investigating the relevance of intact 5-hydroxytryptamine (5-HT) function to the mechanism of anti-OC drug action. The validity of TS-spectrum OCD as a distinct subtype is assessed using a detailed clinical, family, drug treatment response profile in adult OCD patients.

In Study I, patients are divided prospectively into 2 putative subtypes (TS-spectrum and non-TS-spectrum OCD) on the basis of clinical history and direct, structured interviews of family members (approximately 400 interviews).

In Study II, patients enter an 8-week single-blind trial with the potent and selective 5-HT reuptake inhibitor fluoxetine (FX). Patients with an incomplete response to FX alone (approximately 64 patients) are randomized to a 4-week double-blind trial of FX in combination with the dopamine (DA) 2 antagonist olanzapine (OLA) or placebo (PLA).

ELIGIBILITY:
Inclusion criteria required that subjects, ages 14-70 years, have at least a 1-year duration of a current Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) principal diagnosis of OCD. Furthermore, the OCD had to be defined by a rating of "moderate" or greater on the global severity item of the Clinical Global Impressions (CGI) scale and have a Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score of 19 or greater.

Exclusion criteria included primary depression, schizophrenia, or other psychotic disorders; active bipolar disorder; abuse of alcohol or other significant substance within 6 months; increased risk of seizures or history of neurosurgery, encephalitis, or significant head trauma; or a significant medical condition, such as heart, liver, or renal disease. Subjects with an intelligence quotient of less than 80 as determined with the Kaufman Brief Intelligence Test (Kaufman and Kaufman 1990) were excluded.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 1992-09; Primary Completion 2003-01 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
25% reduction in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score from baseline | Baseline, Week s 1, 2, 4, 6, 8, 10, 12, and 14

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Goodman, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Psychiatric Specialty Clinic, Shands Hospital at the University of Florida, Gainesville, Florida
  - University of Florida Behavioral Health Mandarin Clinic, Jacksonville, Florida

REFERENCES:
- [Background] Shapira NA, Ward HE, Mandoki M, Murphy TK, Yang MC, Blier P, Goodman WK. A double-blind, placebo-controlled trial of olanzapine addition in fluoxetine-refractory obsessive-compulsive disorder. Biol Psychiatry. 2004 Mar 1;55(5):553-5. doi: 10.1016/j.biopsych.2003.11.010. PMID 15023585
- [Derived] Koran LM, Bromberg D, Hornfeldt CS, Shepski JC, Wang S, Hollander E. Extended-release fluvoxamine and improvements in quality of life in patients with obsessive-compulsive disorder. Compr Psychiatry. 2010 Jul-Aug;51(4):373-9. doi: 10.1016/j.comppsych.2009.10.001. Epub 2009 Dec 21. PMID 20579510